CLINICAL TRIAL: NCT02385500
Title: Randomized Cross-Over Study of Fesoterodine on Urgency Episodes in Parkinson's Disease Population
Brief Title: Fesoterodine on Urgency Episodes in Parkinson's Disease Population
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient or untimely patient recruitment
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Lysanne Campeau, MDCM, PhD, FRCSC, Assistant Professor, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-007
Record Dates: First submitted 2015-03-04; First posted 2015-03-11 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Urinary Bladder, Overactive; Parkinson Disease
MeSH Terms: conditions — Urinary Bladder, Overactive; Parkinson Disease | interventions — fesoterodine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be started on placebo tablets, similar to fesoterodine 4 mg, and will have the option to escalate as well.
  Interventions: Drug: Fesoterodine; Drug: Placebo
- Fesoterodine (Experimental): Drug intervention of fesoterodine 4 mg once a day in the morning after the two-week washout period. They will have the option to escalate to 8 mg (2 tablets of 4 mg each) after 4 weeks on fesoterodine. Patients will have the option to go back to one tablet (i.e., 4 mg) at any time in the study.
  Interventions: Drug: Fesoterodine; Drug: Placebo

INTERVENTIONS:
Drug: Fesoterodine — For each phase of the study, the participants will receive a total of 84 pills of fesoterodine 4 mg. The study medication will be provided by Pfizer.
  For blinded distribution, each bottle of medications will be labeled with a random number for identification. The participant will indicate in a journal the dose taken each day.
  The study participants will be monitored every 2 weeks with phone calls to assess tolerance or side-effects to the medication.
  Other Names: Toviaz
Drug: Placebo — For each phase of the study, the participants will receive a total of 84 placebo pills. The study medication will be provided by Pfizer.
  For blinded distribution, each bottle of medications will be labeled with a random number for identification. The participant will indicate in a journal the dose taken each day.
  The study participants will be monitored every 2 weeks with phone calls to assess tolerance or side-effects to the medication.
  Other Names: Sugar pill

SUMMARY:
Parkinson's disease (PD) causes several non-motor autonomic symptoms including lower urinary tract dysfunction. Their symptoms can be managed with antimuscarinics with variable efficacy. Fesoterodine offers a new therapeutic molecule to target the symptoms of urinary frequency, urgency and nocturia in this patient population. The purpose of this protocol is to compare the impact of fesoterodine to placebo on urinary urgency and nocturnal sleep problems in a heterogeneous population of PD patients in a cross-over fashion.

A representative number of patients with baseline overactive bladder (OAB) symptoms and Parkinson's disease will be recruited to receive either the active drug or placebo for the first phase of eight weeks. The groups will then be crossed-over during the second phase of eight weeks. The main outcomes assessed will be the urgency episodes on a 3-day voiding diary, as well as the nocturnal sleep problems will be the Parkinson's Disease Sleep Scale (PDSS).

DETAILED DESCRIPTION:
Study purpose and rationale:

Patients with Parkinson's disease (PD) commonly develop lower urinary tract symptoms as their disease severity progresses. The most frequent symptoms are nocturia (night time urinary frequency), urinary frequency and urgency. (1) The effects on voiding function of levodopa and dopamine agonists for the treatment of motor symptoms in patients with PD are not clearly understood because studies conclude conflicting results. (2) Their overactive bladder (OAB) symptoms are primarily managed with antimuscarinics with variable efficacy, and there is concern for possible heightened central side-effects such as cognitive or motor deterioration in this patient population. (3, 4) Current standard of care for PD patients with lower urinary tract symptoms requires a full evaluation with history and physical exam. This is followed by a microscopic urinalysis, a 3-day bladder diary along with several questionnaires. According to their symptoms, some patients may require a non-invasive uroflowmetry and assessment of post void residual, while others will undergo a full urodynamic studies. Management of their voiding symptoms will require initial conservative measures and behavioral modifications (reducing caffeinated drinks and smoking cessation, optimizing fluid intake, weight loss) and bladder training. If this fails to improve their symptoms, oral pharmacotherapy will be offered with antimuscarinics or beta-3 agonists.

The purpose of this protocol is to compare the impact of fesoterodine to placebo on urinary urgency and nocturnal sleep problems in a heterogeneous population of PD patients in a cross-over fashion. Although OAB can be effectively treated, there is compelling and scientifically sound methodological reasons for its use as participants in the study will not face additional risks of serious or irreversible harm from exposure to placebo. Placebo controlled trials are the most rigorous test of treatment efficacy for evaluating a medical therapy and will require fewer subjects than active control trials. Lastly, anticholinergic studies have shown to have a very large placebo effect and are only partially effective in treating voiding symptoms, which justifies the use of a placebo arm.

Sample size:

This is an initial pilot study to identify the effect size of fesoterodine treatment on urgency episodes in patients with PD.

Subjects will be randomized in both groups by stratifying them according to their age group (younger or older than 75 years-old) and gender.

Power analysis and sample size calculation are not relevant in this study given its exploratory nature. The investigators expect to recruit a total of 60 patients to complete the cross-over study for analysis purposes. This number is based on similar design studies, particularly one by Wagg et al. looking at the effects of solifenacin and oxybutynin in older adults with mild cognitive impairment (6). Many other similar studies with groups of subjects varying between 40 and 77 have demonstrated efficacy differences of anticholinergics in a cross-over fashion (7-9).

Design and description of methodology:

This randomized, double-blind, placebo-controlled, crossover, parallel-group study will be carried out in an outpatient clinic. Subjects are assessed and included in the study if they are willing to participate and fit the criteria at Visit 0. They are then randomized to group A or B and undergo a baseline evaluation. Both groups undergo a two-week washout period during which they are given placebo.

Group A subjects will be started on fesoterodine 4 mg once a day in the morning after the two-week washout period. They will have the option to escalate to 8 mg (2 tablets of 4 mg each) after 4 weeks on fesoterodine. Patients will have the option to go back to one tablet (i.e., 4 mg) at any time in the study. At 10 weeks (2 weeks washout and 8 weeks of study tablets), subjects are assessed in the clinic (Visit 1).

Group B subjects will be started on placebo tablets, similar to fesoterodine 4 mg, and will have the option to escalate as well.

All subjects then have a 2-week washout period. After the washout period, subjects will be crossed over to the opposite arm in which the same patterns of outcome assessment and dose titration were maintained. The study will conclude at 20 weeks. At the end of 20 weeks (Visit 2), the investigators' subjects will be interviewed about any side effects, vital signs will be examined, adverse reactions or events monitored, and outcome measures will be documented. Throughout the study, the subjects will be able to drop out anytime with instructions to inform us of their decision and about any adverse effects. Overall, each subject will have 3 clinical visits after enrollment in the study.

Data analysis plan:

The comparison between the 2 arms of the study, the group that initially received fesoterodine with the one that received placebo, will be conducted using chi-square analysis. A 2-sample t test will be used to compare baseline scores between the 2 groups. The Wilcoxon rank-sum test will be used to calculate whether the mean difference of all the outcome measures between treatment and placebo periods is significant.

Differences between placebo and treatments will be adjusted by baseline measures (where available and a 1-sample sign rank tested that the mean difference equated to 0). Any difference will be analyzed as a change from the baseline.

The primary outcome measure will be the number of urgency episodes, with a P value less than .05 considered statistically significant. The present statistical analysis of secondary measures encompasses a number of formal comparisons, and thus a group-wise type I error could occur.

Recruitment procedures:

Study investigators will send a letter to colleagues asking for referrals of eligible patients interested in the study. The study investigators may provide the referring physicians an information sheet about the study to give to the patients. If interested, the patient will contact the investigator. Or, with documented permission from the patient (e.g., note in medical record indicates primary care provider spoke with patient who agreed to be contacted), the investigaor may be allowed to contact patients about enrollment.

Clinics maintain a separate CHR-approved recruitment protocol that asks patients if they will agree ahead of time to be contacted for research. Investigators contact patients about the study in accord with their signed consent. The investigators will consider recruitment when patients with PD present to their clinic with urination symptoms. They will be presented with the option and if they agree, they will then be assessed for inclusion. The investigators will be blinded to the treatment group.

Details on confidentiality:

All data will remain confidential and will be available for access by the investigators only. All records will be identified with a unique identifier, corresponding to the subjects, to maintain confidentiality. Records will be kept in one safe and locked location, and electronic records will be password protected. The study information will be kept for duration of 25 years.

As this is an investigator-initiated trial, Pfizer Canada's role is restricted to providing the medications and placebo, as well as the budget required to do the study. They have approved the current protocol, and will not be involved in further decision-making or data analysis. There are no other potential conflicts of interest.

Statement on ethical considerations:

The study will be conducted according to ethical principles stated in the Declaration of Helsinki (2013), ethics approval will be obtained before initiating study-related procedures, consent forms will take into consideration the well-being, free-will and respect of the participants, including respect of privacy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-85 years-old
* self-reported OAB symptoms for ≥3 months
* a mean of ≥8 micturitions/ 24 hr
* ≥3 urgency episodes/24 hr on a 3-day bladder diary
* at least "some moderate problems" on the Patient Perception of Bladder Condition (PPBC)
* Montreal cognitive assessment (MOCA) score ≥24
* Stable dose of dopaminergic medications and levodopa (between 300 and 1200 mg daily)

Exclusion Criteria:

* Urinary retention: PVR >150 ml (as assessed by bladder scan)
* Contra-indications to fesoterodine
* Unwilling to stop current antimuscarinics
* Patients on anticholinergics for motor disturbances
* Dementia based on clinical evaluation
* Atypical Parkinsonian syndrome
* Deep brain stimulation
* Presence of hallucination

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Urgency episodes | 10 weeks and 20 weeks
  Mean change from baseline in number of urgency episodes per 24 hours

SECONDARY OUTCOMES:
Micturitions | 10 weeks and 20 weeks
  Mean change from baseline per 24 hours in number of micturitions
Urgency urinary incontinence episodes | 10 weeks and 20 weeks
  Mean change from baseline per 24 hours in number of urgency urinary incontinence episodes
Severe urgency episodes | 10 weeks and 20 weeks
  Mean change from baseline per 24 hours in number of severe urgency episodes
Nocturnal micturitions | 10 weeks and 20 weeks
  Mean change from baseline per 24 hours in number of nocturnal micturitions
Incontinence pads used | 10 weeks and 20 weeks
  Mean change from baseline per 24 hours in number of incontinence pads used
Patient's severity of overactive bladder symptoms as measured by OAB-Q score | 10 weeks and 20 weeks
  Mean change from baseline in OAB-Q score
Patient's perception of his bladder condition as measured by PPBC score | 10 weeks and 20 weeks
  Mean change from baseline in PPBC score
Patient's urgency perception as measured by the UPS score | 10 weeks and 20 weeks
  Mean change from baseline in UPS score
Cognitive ability as measured by the MOCA score | 10 weeks and 20 weeks
  Mean change from baseline in MOCA score
Nocturnal sleep disturbances measured by Parkinson's Disease Sleep Scale | 10 weeks and 20 weeks
  Mean change from baseline in PDSS score (on 120)
Safety of fesoterodine in Parkinson's Disease population | 10 weeks and 20 weeks
  Adverse events or reactions

CONTACTS AND LOCATIONS:
Overall Officials: Lysanne Campeau, MD, PhD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winge K, Skau AM, Stimpel H, Nielsen KK, Werdelin L. Prevalence of bladder dysfunction in Parkinsons disease. Neurourol Urodyn. 2006;25(2):116-22. doi: 10.1002/nau.20193. PMID 16402391
- [Background] Campeau L, Soler R, Andersson KE. Bladder dysfunction and parkinsonism: current pathophysiological understanding and management strategies. Curr Urol Rep. 2011 Dec;12(6):396-403. doi: 10.1007/s11934-011-0219-8. PMID 21986769
- [Background] Katzenschlager R, Sampaio C, Costa J, Lees A. Anticholinergics for symptomatic management of Parkinson's disease. Cochrane Database Syst Rev. 2003;2002(2):CD003735. doi: 10.1002/14651858.CD003735. PMID 12804486
- [Background] Donnellan CA, Fook L, McDonald P, Playfer JR. Oxybutynin and cognitive dysfunction. BMJ. 1997 Nov 22;315(7119):1363-4. doi: 10.1136/bmj.315.7119.1363. No abstract available. PMID 9402781
- [Background] Hoyles K, Sharma JC. Olfactory loss as a supporting feature in the diagnosis of Parkinson's disease: a pragmatic approach. J Neurol. 2013 Dec;260(12):2951-8. doi: 10.1007/s00415-013-6848-8. Epub 2013 Feb 3. PMID 23377435
- [Background] Wagg A, Dale M, Tretter R, Stow B, Compion G. Randomised, multicentre, placebo-controlled, double-blind crossover study investigating the effect of solifenacin and oxybutynin in elderly people with mild cognitive impairment: the SENIOR study. Eur Urol. 2013 Jul;64(1):74-81. doi: 10.1016/j.eururo.2013.01.002. Epub 2013 Jan 11. PMID 23332882
- [Background] Abrams P, Cardozo L, Chapple C, Serdarevic D, Hargreaves K, Khullar V; 1032 Study Group. Comparison of the efficacy, safety, and tolerability of propiverine and oxybutynin for the treatment of overactive bladder syndrome. Int J Urol. 2006 Jun;13(6):692-8. doi: 10.1111/j.1442-2042.2006.01387.x. PMID 16834644
- [Background] Zinner N, Tuttle J, Marks L. Efficacy and tolerability of darifenacin, a muscarinic M3 selective receptor antagonist (M3 SRA), compared with oxybutynin in the treatment of patients with overactive bladder. World J Urol. 2005 Sep;23(4):248-52. doi: 10.1007/s00345-005-0507-3. Epub 2005 Nov 8. PMID 16096831
- [Background] Vecchioli-Scaldazza C, Morosetti C, Berouz A, Giannubilo W, Ferrara V. Solifenacin succinate versus percutaneous tibial nerve stimulation in women with overactive bladder syndrome: results of a randomized controlled crossover study. Gynecol Obstet Invest. 2013;75(4):230-4. doi: 10.1159/000350216. Epub 2013 Mar 28. PMID 23548260
- [Background] Chaudhuri KR, Pal S, DiMarco A, Whately-Smith C, Bridgman K, Mathew R, Pezzela FR, Forbes A, Hogl B, Trenkwalder C. The Parkinson's disease sleep scale: a new instrument for assessing sleep and nocturnal disability in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2002 Dec;73(6):629-35. doi: 10.1136/jnnp.73.6.629. PMID 12438461
- [Background] Ginsberg D, Schneider T, Kelleher C, Van Kerrebroeck P, Swift S, Creanga D, Martire DL. Efficacy of fesoterodine compared with extended-release tolterodine in men and women with overactive bladder. BJU Int. 2013 Aug;112(3):373-85. doi: 10.1111/bju.12174. PMID 23826844
- [Background] Coyne KS, Matza LS, Kopp Z, Abrams P. The validation of the patient perception of bladder condition (PPBC): a single-item global measure for patients with overactive bladder. Eur Urol. 2006 Jun;49(6):1079-86. doi: 10.1016/j.eururo.2006.01.007. Epub 2006 Jan 24. PMID 16460875
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- [Background] Cardozo L, Coyne KS, Versi E. Validation of the urgency perception scale. BJU Int. 2005 Mar;95(4):591-6. doi: 10.1111/j.1464-410X.2005.05345.x. PMID 15705086